CLINICAL TRIAL: NCT02829996
Title: Phase II, Randomized, Double-masked, Active-controlled Study of Fixed-Dose Combinations of Trabodenoson and Latanoprost in Subjects With Ocular Hypertension or Primary Open-Angle Glaucoma
Brief Title: Study of Fixed-Dose Combinations of Trabodenoson and Latanoprost in Adults With OHT or POAG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inotek Pharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPC-02-2015
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Results first posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-01

CONDITIONS: Primary Open-Angle Glaucoma (POAG); Ocular Hypertension (OHT)
Keywords: glaucoma; primary open-angle glaucoma; ocular hypertension; adenosine agonist; eye drop; trabodenoson; trabecular meshwork
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — trabodenoson; Latanoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- trabodenoson 6.0% /latanoprost 0.005% QD (Experimental): trabodenoson 6.0% / latanoprost 0.005% QD FDC
  Interventions: Drug: trabodenoson 6.0% / latanoprost 0.005% QD
- trabodenoson 3.0% /latanoprost 0.005% QD (Experimental): trabodenoson 3.0% / latanoprost 0.005% QD FDC
  Interventions: Drug: trabodenoson 3.0% / latanoprost 0.005% QD
- trabodenoson 6.0% /latanoprost 0.0025%QD (Experimental): trabodenoson 6.0% /latanoprost 0.0025% QD FDC
  Interventions: Drug: trabodenoson 6.0% / latanoprost 0.0025% QD
- latanoprost 0.005% QD (Active Comparator): latanoprost 0.005% ophthalmic solution QD
  Interventions: Drug: latanoprost 0.005% QD
- latanoprost 0.0025% QD (Active Comparator): latanoprost 0.0025% ophthalmic solution QD
  Interventions: Drug: latanoprost 0.0025% QD

INTERVENTIONS:
Drug: trabodenoson 6.0% / latanoprost 0.005% QD — Trabodenoson 6.0% / latanoprost 0.005% administered once per day in both eyes and placebo administered once per day in both eyes, for 8 weeks.
  Arms: trabodenoson 6.0% /latanoprost 0.005% QD
Drug: trabodenoson 3.0% / latanoprost 0.005% QD — Trabodenoson 3.0% / latanoprost 0.005% administered once per day in both eyes and placebo administered once per day in both eyes, for 8 weeks.
  Arms: trabodenoson 3.0% /latanoprost 0.005% QD
Drug: trabodenoson 6.0% / latanoprost 0.0025% QD — Trabodenoson 6.0% / latanoprost 0.0025% administered once per day in both eyes and placebo administered once per day in both eyes, for 8 weeks.
  Arms: trabodenoson 6.0% /latanoprost 0.0025%QD
Drug: latanoprost 0.005% QD — Latanoprost 0.005% administered once per day in both eyes and placebo administered once per day in both eyes, for 8 weeks.
  Arms: latanoprost 0.005% QD
Drug: latanoprost 0.0025% QD — Latanoprost 0.0025% administered once per day in both eyes and placebo administered once per day in both eyes, for 8 weeks.
  Arms: latanoprost 0.0025% QD

SUMMARY:
Phase II, randomized, double-masked study to evaluate the efficacy and tolerability of topical ocular delivery of fixed-dosed combinations of trabodenoson and latanoprost in subjects with Ocular Hypertension or Primary Open-Angle Glaucoma.

All subjects who meet the study's enrollment criteria following Screening will undergo washout of all prohibited medications (if washout is needed), including their routine glaucoma medications. During the Placebo Run-In Period, placebo is applied twice daily to both eyes in all subjects. During the Treatment Period, study drug is applied to both eyes for a total of 8 weeks. Each subject will be assigned 4 weeks of AM and 4 weeks of PM dosing in a masked manner. AM vs PM dosing is masked utilizing Placebo in addition to the active drug product. During the Treatment Period, study drug (Active and Placebo) eye drop applications will occur twice daily, in the morning and in the evening. The Treatment Period will be followed by an Observation Period of approximately 7 days wherein no study eye drops are instilled.

The purpose of the study is to assess the overall benefit/risk profile of binocular topical application of different doses of trabodenoson (3.0% and 6.0%) when combined with latanoprost (0.005% or 0.0025%) one drop daily (QD) for 8 weeks.

DETAILED DESCRIPTION:
This is a phase II, randomized, double-masked study to evaluate the efficacy and tolerability of topical ocular delivery of fixed-dose combinations of trabodenoson and latanoprost in subjects with OHT or POAG.

The Primary Objective of this Trial is to evaluate the efficacy of different topical ocular doses of trabodenoson (3.0% and 6.0%) when added to latanoprost (0.005% or 0.0025%), one drop daily to both eyes over two consecutive 4 week periods. The Secondary Objective is to evaluate the tolerability and safety of different doses of trabodenoson (3.0% and 6.0%) when added to latanoprost (0.005% or 0.0025%), one drop daily to both eyes over two consecutive 4 week periods. the Hypotheses is that topical ocular co-administration of 3.0% or 6.0% trabodenoson plus latanoprost 0.0025% or 0.005% ophthalmic formulation will reduce IOP and be well-tolerated.

All subjects who meet the study's enrollment criteria following Screening will undergo washout of all prohibited medications, including their routine glaucoma medications. During the Placebo Run-In Period, placebo (vehicle control matched to trabodenoson) is applied twice daily to both eyes in all subjects. During the Treatment Period, study drug is applied to both eyes for a total of 8 weeks. Each subject will be assigned 4 weeks of AM and 4 weeks of PM dosing in a manner that is masked to the patient. The Treatment Period will be followed by an Observation Period of approximately 7 days wherein no study eye drops are instilled.

To mimic what is generally seen in clinical trials, the number of subjects with ocular hypertension as their diagnosis will be limited to approximately 30% of the total subjects enrolled. Additionally, so the trial mirrors the general population demographics (so as to improve generalizability of the results) the proportion of African American subjects will be approximately 25% or less but not less than 12% of the total subjects enrolled.

The purpose of the study is to assess the efficacy, tolerability, and safety of binocular topical application of different doses of trabodenoson (3.0% and 6.0%) when added to latanoprost (0.005% or 0.0025%) one drop daily over two consecutive 4 week periods in subjects with POAG or OHT. Data collection will include efficacy (masked-IOPs), local (ophthalmic) and systemic tolerability and safety assessments

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ocular hypertension (OHT) or primary open-angle glaucoma (POAG)
* Mean Intraocular pressure (IOP) of ≥25 and ≤34

Exclusion Criteria:

* Significant visual field loss or any new field loss within the past year
* Cup-to-disc ratio >0.8
* Central corneal thickness <490 µm or >610 µm
* A recent (acute) or chronic medical condition that might obfuscate the Subject's study data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2016-08-19 (Actual); Primary Completion 2017-05-24 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cadmus C Rich, MD,MBA,CPE, Study Director — Inotek Pharmaceuticals Corp.
Locations (1):
- Inotek Pharmaceuticals Corporation, Lexington, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Trabodenoson 6.0% / Latanoprost 0.005% QD: trabodenoson 6.0% / latanoprost 0.005% Fixed-Dose Combination
  trabodenoson 6.0% / latanoprost 0.005% QD: Trabodenoson 6.0% / latanoprost 0.005% administered once per day in both eyes and placebo administered once per day in both eyes, for 8 weeks.
- Trabodenoson 3.0% / Latanoprost 0.005% QD: trabodenoson 3.0% / latanoprost 0.005% Fixed-Dose Combination
  trabodenoson 3.0% / latanoprost 0.005% QD: Trabodenoson 3.0% / latanoprost 0.005% administered once per day in both eyes and placebo administered once per day in both eyes, for 8 weeks.
- Trabodenoson 6.0% / Latanoprost 0.0025% QD: trabodenoson 6.0% / latanoprost 0.0025% Fixed-Dose Combination
  trabodenoson 6.0% / latanoprost 0.0025% QD: Trabodenoson 6.0% / latanoprost 0.0025% administered once per day in both eyes and placebo administered once per day in both eyes, for 8 weeks.
- Latanoprost 0.005% QD: latanoprost 0.005% ophthalmic solution
  latanoprost 0.005% QD: Latanoprost 0.005% administered once per day in both eyes and placebo administered once per day in both eyes, for 8 weeks.
- Latanoprost 0.0025% QD: latanoprost 0.0025% ophthalmic solution
  latanoprost 0.0025% QD: Latanoprost 0.0025% administered once per day in both eyes and placebo administered once per day in both eyes, for 8 weeks.
Period: Overall Study
Arm/Group | Trabodenoson 6.0% / Latanoprost 0.005% QD | Trabodenoson 3.0% / Latanoprost 0.005% QD | Trabodenoson 6.0% / Latanoprost 0.0025% QD | Latanoprost 0.005% QD | Latanoprost 0.0025% QD
Started | 39 | 39 | 40 | 41 | 42
Completed | 38 | 39 | 40 | 41 | 42
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trabodenoson 6.0% / Latanoprost 0.005% QD | Trabodenoson 3.0% / Latanoprost 0.005% QD | Trabodenoson 6.0% / Latanoprost 0.0025% QD | Latanoprost 0.005% QD | Latanoprost 0.0025% QD | Total
Number analyzed (Participants) | 39 | 39 | 40 | 41 | 42 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (12.08) | 64.4 (9.18) | 68.8 (8.43) | 66.5 (9.84) | 66.4 (8.57) | 66.0 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 23 | 19 | 22 | 27 | 108
  Male | 22 | 16 | 21 | 19 | 15 | 93
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 1 | 2 | 1 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 9 | 8 | 9 | 10 | 44
  White | 30 | 27 | 31 | 32 | 32 | 152
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 39 | 39 | 40 | 41 | 42 | 201
Baseline IOP [Mean (Standard Deviation); unit: mm of mercury] — mm of mercury on Goldmann Applanation Tonometry
  mm of mercury | 27.67 (2.329) | 27.17 (2.278) | 27.28 (2.155) | 27.48 (2.627) | 27.31 (2.276) | 27.38 (2.323)

OUTCOME MEASURES:

1. Primary Outcome: Mean Intraocular Pressure (IOP)
Description: Daily change from diurnal baseline in IOP
Time Frame: Two Months
Population: Intent to treat
Measure: Mean (Standard Error); unit: mm of mercury
Arm/Group | Trabodenoson 6.0% / Latanoprost 0.005% QD | Trabodenoson 3.0% / Latanoprost 0.005% QD | Trabodenoson 6.0% / Latanoprost 0.0025% QD | Latanoprost 0.005% QD | Latanoprost 0.0025% QD
Number analyzed (Participants) | 39 | 39 | 40 | 41 | 42
mm of mercury | -6.4 (0.48) | -6.8 (0.56) | -6.4 (0.56) | -7.1 (0.46) | -5.9 (0.53)

2. Other Pre Specified Outcome: Safety Parameters, Including Treatment Emergent Adverse Events, to Assess Tolerability and Safety.
Description: Collection of safety parameters, including treatment emergent adverse events, laboratory assessments, to assess tolerability and safety.
Time Frame: Through Study Completion, up to 9 weeks.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Trabodenoson 6.0% / Latanoprost 0.005% QD | Trabodenoson 3.0% / Latanoprost 0.005% QD | Trabodenoson 6.0% / Latanoprost 0.0025% QD | Latanoprost 0.005% QD | Latanoprost 0.0025% QD
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39 | 0/40 | 0/41 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39 | 0/40 | 0/41 | 0/42
Other Adverse Events (participants affected / at risk) | 9/39 | 5/39 | 6/40 | 3/41 | 5/42
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trabodenoson 6.0% / Latanoprost 0.005% QD (N=39) | Trabodenoson 3.0% / Latanoprost 0.005% QD (N=39) | Trabodenoson 6.0% / Latanoprost 0.0025% QD (N=40) | Latanoprost 0.005% QD (N=41) | Latanoprost 0.0025% QD (N=42)
UTI (Infections and infestations) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (2)
Eye Discharge (Eye disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival Hyperaemia (Eye disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Punctate Keratitis (Eye disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/96/NCT02829996/SAP_000.pdf
  • Study Protocol (2016-06-26): https://cdn.clinicaltrials.gov/large-docs/96/NCT02829996/Prot_001.pdf